CLINICAL TRIAL: NCT06377514
Title: Clinical Investigation of the TECNIS® Next-Generation Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PCOL109PHNG
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Test IOL (Experimental): DEN00V
  Interventions: Device: Test IOL Model DEN00V
- Control IOL (Active Comparator): DCB00
  Interventions: Device: Control IOL Model DCB00

INTERVENTIONS:
Device: Test IOL Model DEN00V — Eligible subjects will be randomized in a 1:1 ratio to receive the Test IOL Model DEN00V in both eyes for the duration of the study
  Arms: Test IOL
Device: Control IOL Model DCB00 — Eligible subjects will be randomized in a 1:1 ratio to receive the control IOL Model DCB00 in both eyes for the duration of the study
  Arms: Control IOL

SUMMARY:
Prospective, multicenter, bilateral, interventional, controlled, masked (sponsor, subjects, and evaluators), randomized clinical trial.

ELIGIBILITY:
INCLUSION CRITERIA

To be considered for enrollment in this study, patient must:

* be at least 22 years old
* have cataracts in both eyes
* sign the written informed consent
* be willing and able to comply with examination procedures
* understand, read and write English to complete informed consent and questionnaires
* be available for study follow-up visits EXCLUSION CRITERIA

Patient will not be eligible to take part in the study if:

* currently participating in any other clinical study or have participated in a clinical study during the last 30 days
* have a certain disease/illness, such as poorly controlled diabetes
* have certain ocular conditions, such as uncontrolled pressure in the eye
* taking medication that may affect vision
* pregnant, plan to become pregnant during the study, or are breastfeeding

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Monocular photopic DCIVA (first eyes) at 66 cm | 6 months
  Mean DCIVA (logMAR) in test lens group is statistically significantly better (smaller) than in the control lens group
Monocular Depth of Focus | 6 months
  Monocular depth of defocus where visual acuity is 0.20 logMAR or better (measured only negative direction from zero) for first eyes at 6 months
Monocular Photopic BCDVA at 4m | 6 months
  Monocular photopic BCDVA at 4 meters for first eyes at 6 months
Monocular Photopic DCVA at 100 cm | 6 months
  Monocular photopic DCVA at 100 cm for first eyes at 6 months

SECONDARY OUTCOMES:
Monocular photopic DCNVA at 40 cm (first eyes) | 6 months
  Mean DCNVA (logMAR) in the test lens group is statistically significantly better (smaller) than in the control lens group

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision, Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (9):
- United States (9):
  - Empire Eye & Laser Center, Bakersfield, California
  - Levenson Eye Associates, Jacksonville, Florida
  - Jones Eye Center, Sioux City, Iowa
  - OCLI Vision, Garden City, New York
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Berkeley Eye Institute, Houston, Texas
  - Whitsett Vision Group, Houston, Texas
  - Parkhurst NuVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu